CLINICAL TRIAL: NCT02924363
Title: Effect of MitraClip on Reverse Cardiac Remodeling Assessed by CMR and Echocardiography: The MITRA-REVERSE Study A Prospective Multicenter Study
Brief Title: Effect of MitraClip on Acute and Chronic Reverse Cardiac Remodeling Assessed by CMR: The MITRA-REVERSE Study
Acronym: MITRA-REV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dipan Shah (Other)
Collaborators: Piedmont Heart Institute, Inc., Atlanta, GA (Industry)
Responsible Party: Sponsor-Investigator, Dipan Shah, Dipan J. Shah, MD, Director Cardiovascular MRI Laboratory, Houston Methodist DeBakey Heart & Vascular Center (HMDHVC), The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00013041
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Mitral Regurgitation
Keywords: Cardiac Magnetic Resonance; Mitra Clip; Mitral Valve
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Blood Specimen Collection; Phlebotomy; Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimen will be stored for subsequent biomarker testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm (cardiac MRI & hematocrit blood sample): Patients will undergo a pre- & post- MitraClip procedure cardiac magnetic resonance imaging (CMR) scan with an FDA cleared MRI scanner and with or without an FDA approved contrast dye. The scan and the blood draw to assess the hematocrit is research, the MitraClip procedure is standard of care for these patients.
  Interventions: Diagnostic Test: Cardiac MRI with or without contrast dye; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Cardiac MRI with or without contrast dye — MRI scans of the heart are performed before and after the MitraClip clinical procedure with an FDA cleared device with or without an FDA approved contrast dye.
Diagnostic Test: Blood sample — Blood samples collected to calculate hematocrit for measurements of the CMR extracellular matrix.
  Other Names: phlebotomy, Complete Blood Count (CBC) for hematocrit value

SUMMARY:
The purpose of this study is to use cardiac magnetic resonance (CMR) and echocardiography to define the anatomic and functional remodeling that results from MitraClip implantation. A total of sixty (60) patients undergoing MitraClip implantation will be enrolled across multiple sites. The severity of mitral regurgitation, cardiac morphology and function will be assessed in these patients by taking cardiac magnetic resonance imaging with an FDA approved contrast agent at BASELINE (within 30 days prior to MitraClip implantation), during the ACUTE REMODELING PHASE (pre-discharge following implantation), and during the CHRONIC REMODELING PHASE (6 months post-implantation).

DETAILED DESCRIPTION:
Percutaneous mitral valve repair is expanding treatment options for patients suffering from symptomatic mitral regurgitation (MR). The overall objective of the procedure is to reduce the degree of MR, which may lead to improvement in: 1) hemodynamics, an increase in systemic stroke volume and decrease in left atrial (LA) pressure; 2) left ventricular (LV) and LA volumes (reverse remodeling); and 3) efficiency in LV mechanics (decreased wall stress and improved fluid kinetics in the LV). The MitraClip System is the only percutaneous therapy available for high surgical risk patients with significant MR (Figure 1). Two-dimensional Echocardiography (2-D) data from the Endovascular valve edge-to-edge study (EVEREST trial) showed reverse modeling of LA and LV volumes in patients with primary MR after MitraClip implantation. In a separate study, patients with secondary MR who were non-respondent to cardiac resynchronization therapy (CRT) demonstrated improvement in LA and LV volumes post-MitraClip implantation [3]. Two smaller studies have also demonstrated the feasibility of using CMR to show improvement in LA and LV volumes post-MitraClip.

Immediate post-procedural reduction in MR or, conversely the degree of residual MR, has been shown to be a predictive factor of long-term improvement in MR, LV and LA reverse remodeling, and survival. Current assessment of MR reduction post-MitraClip relies on a combination of indirect hemodynamic parameters, such as LA pressure and 2-D Echo parameters, which are semi-quantitative at best. Therefore, a rapid and accurate quantitative method to assess the degree of residual MR is of great need to complement other invasive and indirect/qualitative echo parameters. This will not only improve the reliability and reproducibility of residual MR assessment post-Mitraclip, but will also provide an objective index to define successful procedural outcomes. The latter may potentially help in decision making for the placement of additional clips to further reduce MR. Of the quantitative color Doppler parameters used to measure the degree of MR, regurgitant volume/fraction (RV/RF) is probably the most optimal index. The Mitra-clip has been shown to distort data from the flow convergence (PISA) method, resulting in complicated and unreliable assessments of MR. Similarly, vena contracta (VC) is also distorted by the Mitra-Clip, which can lead to unreliable and unreproducible measures of MR. It has been previously shown that real-time volume color flow Doppler (RT-VCFD) trans-thoracic echocardiography (TTE) is useful to quantify RV/RF and comparable to CMR. Since 3-D transesophageal echocardiography is commonly used for Mitra-Clip assessment, the same principle can be applied to RT-VCFD TEE. The preliminary experience with this approach has shown promise.

The attenuation of LV/LA remodeling, defined as the reduction in LV end-systolic volume and LA volume, is an important goal of MR reduction after Mitra-clip placement. Post Mitra-Clip TTE is limited by acoustic windows in at least one-third of patients, rendering 3-D TTE measurements of LV/LA volumes unfeasible. Contrast Echo can mitigate the drawbacks of TTE, but 2-D volumes are under-estimated compared to CMR. Hence, the impact of MR reduction by Mitra-clip on LV/LA remodeling is best determined by CMR. Furthermore, CMR will provide an independent reference standard to validate RV/RF measured by RT-VCFD TEE pre- and post-Mitra-clip placement.

Cardiac morphology and function have primarily been assessed by echocardiography in patients undergoing percutaneous mitral valve repair, which has known limitations with regard to image quality and reproducibility. Transesophageal echocardiogram (TEE) is a standard technique for assessing MR and intra-procedural guidance; however, TEE quantification of MR and effective orifice area after MitraClip placement can be challenging in a double-orifice valve model and has not been well validated. While reduction in chamber size after MitraClip placement has been demonstrated, prior analysis has been limited by imprecise assessment of regurgitation severity resulting in successful remodeling and clinical improvement. Alternatively, CMR is a validated noninvasive technique that could be utilized to evaluate the heart and valve structure, function, and myocardial fibrosis without any geometric assumptions or harmful radiation.

CMR enables noninvasive evaluation of cardiac anatomy, including great arteries and veins, and cardiac chambers. It provides excellent evaluation of both the left ventricle (LV) and right ventricle (RV), including ventricular size, thickness, wall motion, volumes, and ejection fraction (EF), without the need for geometric assumptions. Many consider CMR to be the gold standard for quantifying ventricular volumes and EF. In addition, CMR can better define valvular disease due to its ability to precisely quantify regurgitant volumes and fractions without limitation from acoustic windows, or highly eccentric/multiple jets. Feasibility and safety of CMR after MitraClip placement has previously been shown [5]. In order to obtain a concurrent comparison of CMR with echocardiography, a comprehensive 2D/3D echo with Doppler will be performed immediately before or after the CMR scan. The echocardiography protocol will be outlined in detail in the Echo Imaging Manual.

Additionally, a SUBSTUDY (MITRA-REVERSE FIBROSIS) will explore newer CMR techniques, such as T1 mapping and extracellular volume fraction quantification, can now non-invasively quantify the extent of diffuse extracellular matrix expansion as a surrogate for interstitial fibrosis, and are supported by histological validation. The interplay between diffuse interstitial fibrosis, volume overload reduction (via decrease in mitral regurgitation), and subsequent LV reverse remodeling are not well understood. It is possible that increasing burden of diffuse interstitial fibrosis at baseline may prevent, blunt, or delay the reverse remodeling that occurs following volume overload reduction. Alternatively, volume overload reduction and reverse LV remodeling may lead to subsequent reduction in diffuse interstitial fibrosis A sub-study with gadolinium contrast administration will attempt to address these questions. MR patients without contraindications to gadolinium will be enrolled into the sub-study that includes pre- and post-gadolinium contrast imaging in order to quantifying LV myocardial replacement and interstitial fibrosis, as well as papillary muscle fibrosis. Recently, in a cohort of 48 patients with chronic MR undergoing surgical mitral valve repair, it has been demonstrated that the presence of LV myocardial fibrosis assessed with delayed-enhancement CMR was an independent predictor of increased adverse clinical outcomes. Similarly, in this sub-study it is intended to examine the correlation between the presence and extent of myocardial replacement and interstitial fibrosis to clinical response, as assessed by New York Heart Association (NYHA) class and Kansas City Cardiomyopathy Questionnaire, following a MitraClip procedure. Moreover, a new technique to quantify replacement fibrosis in the papillary muscles may be exploited in the gadolinium sub-study that could provide additional information, as the papillary muscles of the left ventricle are key components of the mitral valve apparatus. Papillary muscles connect the LV wall with the mitral leaflets and annulus, and regulate the location of the mitral leaflets. Thus, the geometry and function of papillary muscles contribute to mitral valve function and an accurate evaluation is key in understanding the pathophysiology of mitral valve disease. This evaluation of the papillary muscles will rely on a new procedure that is based on the use of a novel dark blood delayed enhancement imaging technique.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 years of age or older.
2. Negative pregnancy test (serum or urine β-HCG) within 24 hours of gadolinium contrast administration, if female and of child-bearing potential. In addition, all female patients of childbearing potential must agree to use a medically accepted method of contraception throughout the study (this applies only to patients in the gadolinium sub-study).
3. Symptomatic severe mitral regurgitation (grade 3-4+).
4. Undergoing MitraClip implantation due to increased surgical risk.
5. Patients or legally authorized representatives who have the ability to understand the requirements of the study and provide written consent/assent to participate and agree to abide by the study requirements.

Exclusion Criteria:

1. The patient is enrolled in the Clinical Outcomes Assessment of the MitraClip Percutaneous Therapy Trial (COAPT).
2. The patient is scheduled to undergo percutaneous coronary intervention with MitraClip procedure.
3. The patient has Stage D Congestive Heart Failure or inability to lay flat for 60 minutes.
4. The patient has a medical condition, serious concurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up.
5. The patient has contraindications to CMR, including:

   1. Implanted defibrillator or pacemaker that is not MRI conditional
   2. Epicardial pacemaker leads, or any abandoned leads
   3. Ferromagnetic aneurysm clip
   4. Ferromagnetic halo device
   5. Cochlear implants
   6. Implanted infusion pumps
   7. Severe claustrophobia
   8. Any other conditions which represent contraindication to CMR.
6. The patient is clinically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multicenter, longitudinal observational study to evaluate reverse cardiac remodeling following MitraClip therapy for significant mitral regurgitation. A schematic overview of the study design is shown in Figure 4. Subjects with 3-4+ mitral regurgitation, who are already scheduled to undergo MitraClip therapy, will be enrolled, if they do not meet any of the exclusion criteria. Patients will undergo CMR and echocardiographic assessment of their mitral regurgitation and cardiac morphology/function prior to MitraClip placement. Patients without contraindication to gadolinium will undergo late gadolinium enhancement CMR to assess for LV and papillary muscle replacement fibrosis, and T1 mapping (pre and post contrast) to assess for LV diffuse interstitial fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular remodeling | baseline comparison to 6 month scan
  Serial CMR scans obtained to document changes in the ventricular remodeling

CONTACTS AND LOCATIONS:
Overall Officials: Dipan J Shah, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Piedmont Heart Institute, Atlanta, Georgia
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No